CLINICAL TRIAL: NCT01935167
Title: A Phase Ⅱ, Prospective, 24 Weeks, Double-blind, Placebo-controlled, Randomized, Multi-center Clinical Trial for the Evaluation of the Efficacy and Safety of DW1029M on Microalbuminuria in Patients With Diabetic Nephropathy
Brief Title: To Determine the Efficacy and Safety of DW1029M on Microalbuminuria in Patients With Diabetic Nephropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dong Wha Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DW1029M
Record Dates: First submitted 2013-08-30; First posted 2013-09-04 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: Diabetic Nephropathy
Keywords: Microalbuminuria
MeSH Terms: conditions — Diabetic Nephropathies

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- A Group (Experimental): DW1029M 600mg for 24 weeks
  Interventions: Drug: DW1029M 600mg
- B Group (Experimental): DW1029M 1200mg for 24 weeks
  Interventions: Drug: DW1029M 1200mg
- C Group (Placebo Comparator): Placebo for 24 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DW1029M 600mg — DW1029M 150mg 2 tablets b.i.d
  Other Names: DW1029M 150mg 2 tablets
  Arms: A Group
Drug: DW1029M 1200mg — DW1029M 300mg 2 tablets b.i.d
  Other Names: DW1029M 300mg 4 tablets
  Arms: B Group
Drug: Placebo — Placebo 2 tablets b.i.d.
  Arms: C Group

SUMMARY:
Phase 2 clinical study to evaluate of the efficacy and safety of DW1029M on microalbuminuria in Patients With Diabetic Nephropathy

DETAILED DESCRIPTION:
A Phase Ⅱ, prospective, 24 weeks, double-blind, placebo-controlled, randomized, multi-center clinical trial for the evaluation of the efficacy and safety of DW1029M on microalbuminuria in Patients With Diabetic Nephropathy

ELIGIBILITY:
Inclusion Criteria:

* Has confirmed diabetic mellitus prior to 6years
* Has confirmed microalbuminuria 30 ~ 299㎍/㎎creatinine prior to 5months one time and microalbuminuria 30 ~ 299㎍/㎎creatinine during screening period
* Blood Pressure(BP) ≤ 150 / 90 mmHg
* estimated glomerular filtration rate(eGFR) ≥ 30 ml/min/1.73m2
* Hemoglobin A1c(HbA1c) ≤ 9%
* Low density lipoprotein(LDL-C) ≤ 130mg/dl

Exclusion Criteria:

* kidney or liver disease as follows i.Serum Creatinine > 2.0mg/dl ii.Alanine Aminotransferase(ALT) or Aspartate Aminotransferase(AST) > 2 x Upper Limit Normal(ULN) iii.Total Bilirubin > 2 x ULN
* Organic gastrointestinal disorder or Chronic gastroenterologic disorders prior to 6 months as follows [NOTE] Active Crohn's disease, Active ulcerative colitis, Chronic peptic ulcer disease, etc.
* cardiovascular disease prior to 3 months as follows [NOTE] Unstable angina pectoris, Myocardial infarction, Coronary artery bypass surgery, Percutaneous Transluminal Coronary Angioplasty, transient ischemic attack, cerebrovascular accident etc.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2013-10; Primary Completion 2014-08 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
log ACR | 24 weeks after 1st administration
  logarithm of the Albumin Creatinine Ratio(ACR) after 24 weeks

SECONDARY OUTCOMES:
Log UAE | 24 weeks after 1st administration
  Urinary Albumin Excretion(UAE) after 12 and 24 weeks
eGFR | 12 and 24 weeks after 1st administration
  estimated Glomerular Filtration Rate(eGFR) after 12 and 24 weeks
log ACR | 12 weeks after 1st administration
  logarithm of the Albumin Creatinine Ratio(ACR) after 12 weeks
SCC | 12 and 24 weeks after 1st administration
  Serum Creatinine Concentration(SCC) after 12 and 24 weeks
Cystatin C | 12 and 24 weeks after 1st administration
  Cystatin C after 12 and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: MoonKyu Lee, Professor, Principal Investigator — Samsung Medical Center
Locations (1):
- DongWha Pharm, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No